CLINICAL TRIAL: NCT00005493
Title: Observational Aspirin Use and CVD in the Physicians' Health Study
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5010; R03HL058476 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction; Cerebrovascular Accident
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction; Stroke

SUMMARY:
To analyze existing data from the Physicians Health Study (PHS), a randomized primary prevention trial of low-dose aspirin and beta carotene conducted among 22,071 U.S. male physicians, to address questions concerning aspirin and cardiovascular (CV) disease that could not adequately be addressed during the randomized aspirin period.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

The aspirin component of the trial was terminated on January 25, 1988, due to a demonstrated benefit of aspirin on myocardial infarction. At that time, however, the number of strokes and CV deaths experienced by trial participants was inadequate to definitively evaluate these endpoints. The beta carotene component of the trial continued uninterrupted until its scheduled termination in December, 1996. During this period detailed information continued to be collected on post-trial aspirin use through annual questionnaires. As of October, 1995, the number of deaths, including cardiovascular deaths, had increased fourfold from that in the randomized period, and the number of strokes had increased 3.5 times. The investigators used data from both the randomized aspirin period and the observational period following the trial to assess the impact of aspirin use on cardiovascular and total mortality, and the long-term impact of aspirin use on subsequent stroke and MI. The methods included analyses of both randomized aspirin assignment and of time-varying aspirin use, as assessed on the annual questionnaires. Because of the potential for bias, the propensity for aspirin use, particularly during the observational period was taken into account. Analyses included use of proportional hazards models allowing for both time-varying effects of aspirin use and controlling for time-varying confounders, as well as more complex procedures using causal modeling.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-04; Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Cook — Brigham and Women's Hospital

REFERENCES:
- [Background] Cook NR, Hebert PR, Manson JE, Buring JE, Hennekens CH. Self-selected posttrial aspirin use and subsequent cardiovascular disease and mortality in the physicians' health study. Arch Intern Med. 2000 Apr 10;160(7):921-8. doi: 10.1001/archinte.160.7.921. PMID 10761956
- [Background] Cook NR, Cole SR, Hennekens CH. Use of a marginal structural model to determine the effect of aspirin on cardiovascular mortality in the Physicians' Health Study. Am J Epidemiol. 2002 Jun 1;155(11):1045-53. doi: 10.1093/aje/155.11.1045. PMID 12034583